CLINICAL TRIAL: NCT04871243
Title: Qualitative Study Evaluating Opinions Regarding HPV Vaccinnation in Boys' Parents Aged From 11 to 14 Years Old
Brief Title: Children Vaccination From 11 to 14 Years Old
Acronym: QUALIOPIVAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Eure-Seine (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A00660-41; CHES N°21/01 (Other: CH Eure-Seine)
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Vaccination Refusal; Opinions
Keywords: human papilloma virus; vaccination
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative Interview — Individual semi-structured interviews

SUMMARY:
The human papilloma virus infection is the most frequent sexually transmitted infection around the world. In the vast majority of cases, these are inapparent infections that disappear spontaneously. In some cases, the HPV infection persists and can generate anogenital warts or cancer.

In France, the papillomavirus is responsible for 6000 new cases of cancer/year with several possible localizations : cervical, anal, penile, oropharyngeal, vulvar or vaginal. Among them, 4580 new cases of cancer/year occur in women, and half of them are diagnosis of cervical cancer. A quarter of cancers caused by papillomavirus occur in men.

In France, the commercialization of anti-HPV vaccine in 2007 was addressed only to girls, in order to gain a group immunity that would therefore protect the boys. This vaccination did not achieve the cover immunization target that were announced: the objective was fixed at 60% of vaccination coverage and at the end of 2018, only 24% was achieved on the complete vaccination schedule. In December 2019, the French National Authority for Health recommended the anti-HPV vaccinations in girls and boys.

DETAILED DESCRIPTION:
This qualitative study evaluates parents' opinion regarding the vaccination and the HPV. Parent's eligible to participate in this study are those with boys between 11 and 14 years old.

The anti-HPV vaccination is perceived favorably in 38% of parents, but 42% of parents are undecided.

The investigators would like to evaluate qualitatively the opinions and the obstacles in this vaccination, using interviews in parents of boys aged between 11 and 14 years old.

ELIGIBILITY:
Inclusion Criteria:

* parents having boys between 11 and 14 years old, followed-up by a general practitioner that participate in the study
* signed inform consent form

Exclusion Criteria:

* language barrier that could prevent the understanding or formulation of opinions during the interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients followed-up by a general practitioner that participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of knowledge and understanding of papillomavirus and opinions related to anti-HPV vaccination | 4 months

SECONDARY OUTCOMES:
Concept identification to ameliorate the vaccination coverage by overcoming the obstacles | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- CH Eure-Seine, Évreux, France